CLINICAL TRIAL: NCT00716053
Title: Phase 3 Study of the Biologic Lung Volume Reduction (BLVR) System in Patients With Advanced Upper Lobe Predominant Emphysema
Brief Title: Phase 3 Study of the Biologic Lung Volume Reduction (BLVR) System in Advanced Upper Lobe Predominant (ULP) Emphysema
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Aeris Therapeutics (Industry)
Responsible Party: Program Manager, Clinical Dept.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-C08-001
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2010-01

CONDITIONS: Advanced Upper Lobe Predominant Emphysema
Keywords: emphysema; chronic obstructive pulmonary disease; COPD; lung volume reduction; LVRS; BLVR; Aeris
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BLVR (Experimental)
  Interventions: Drug: BLVR
- Saline (Sham Comparator)
  Interventions: Drug: BLVR

INTERVENTIONS:
Drug: BLVR — BLVR 20 mL

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of the 20 mL BLVR System in treating patients with advanced upper lobe predominant emphysema.

DETAILED DESCRIPTION:
Patients with emphysema currently have limited treatment choices. Many patients are treated with steroids and inhaled medications,which often provide little or no benefit.

In recent years, lung volume reduction surgery has become an accepted therapy for advanced emphysema. Lung volume reduction surgery involves the removal of diseased portions of the lung in order to enable the remaining, healthier portions of the lung to function better. This procedure, although effective for many patients, is complicated and is accompanied by substantial morbidity and mortality risk.

Aeris Therapeutics has developed the Biologic Lung Volume Reduction (BLVR) System to achieve lung volume reduction without surgery and its attendant risks. With BLVR, a physician uses a bronchoscope to direct treatment to the most damaged areas of the patient's lungs. The treatment delivers a precisely proportioned proprietary mixture of drugs and biologics which, when combined at the treatment site, form a bioabsorbable gel. The gel is comprised of clotting proteins that deliver the treatment, an antibiotic to prevent infection and drugs designed to remodel damaged areas of the lungs-actually using the body's natural scar formation response to permanently collapse the diseased areas. This reduction in lung volume creates more space for adjacent healthier parts of the lungs to function more effectively.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-12; Study Completion 2009-12

PRIMARY OUTCOMES:
Improvement in pulmonary function and respiratory symptoms | 6 months

REFERENCES:
- [Background] Ingenito EP, Berger RL, Henderson AC, Reilly JJ, Tsai L, Hoffman A. Bronchoscopic lung volume reduction using tissue engineering principles. Am J Respir Crit Care Med. 2003 Mar 1;167(5):771-8. doi: 10.1164/rccm.200208-842OC. Epub 2002 Oct 11. PMID 12406835
- [Background] Reilly J, Washko G, Pinto-Plata V, Velez E, Kenney L, Berger R, Celli B. Biological lung volume reduction: a new bronchoscopic therapy for advanced emphysema. Chest. 2007 Apr;131(4):1108-13. doi: 10.1378/chest.06-1754. PMID 17426216